CLINICAL TRIAL: NCT03334656
Title: Controlled Comparison of a Traditional Dressing Versus a Biologic Dressing Composed of Fetal Fibroblasts and Keratinocytes in Association With a Collagen Matrix on Skin Donor Sites
Acronym: CICAFAST
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: It was decided to terminate the study prematurely due to insufficient enrolment, despite extensions to the enrolment period.
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: RC16_0019
Record Dates: First submitted 2017-10-30; First posted 2017-11-07 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Split Thickness Skin Graft; Wound Healing
Keywords: Split thickness skin graft donor site; wound healing; Fetal skin bioconstruct; Fibroblasts; Keratinocytes
MeSH Terms: interventions — Biological Dressings

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biological Dressing (Experimental): It is a cellularized dressing of 100 cm² composed of fetal skin cells associated to a bovine collagen matrix:
  * Fetal skin cells were obtained from a single fetal skin sample and consist in two clinical grade banks of keratinocytes (reference BKF07 K CB1) and fibroblasts (reference BKF07 WCB F d P3) produced at the UTCG. These two clinical grade cells banks were fully characterized and secure.
  * The matrix is a customized type I calf collagen produced by the company Symatese. Symatese's collagen is in compliance with the European requirements
  Interventions: Biological: biological dressing
- Paraffin Gauze Dressing (Active Comparator): It is a low-adherent, sterile paraffin Tulle Gras dressing made from open weave gauze. The gauze has interlocking threads which minimize fraying when the dressing is cut to shape. JELONET® dressings are non-medicated and are used as a primary wound contact layer with paraffin present to reduce the adherence of the product to the surface of a granulating wound.
  JELONET® is a product of Smith-Nephew, it has the CE-mark (n°0086) and the class of this medical device is IIa.
  The features of this dressing are: Soft paraffin base, Sterile leno weave presentation, Comprehensive size range.
  Interventions: Other: Paraffin gauze dressing

INTERVENTIONS:
Biological: biological dressing — to test a biological dressing on the wound healing of the split-thickness skin graft donor site
  Arms: Biological Dressing
Other: Paraffin gauze dressing — standard intervention : Paraffin gauze dressing on the wound healing
  Arms: Paraffin Gauze Dressing

SUMMARY:
Cell-based engineered skin substitutes are promising to treat difficult-to-heal acute and chronic wounds such as large/deep burns, ulcers resistant to conventional therapies or surgical wounds. Cultured autologous epidermal cell-based therapy is used for more than two decades as permanent wound coverage for large burns. Although this technique has been shown to improve outcomes in patients with large burn injuries, its clinical use is limited by the creation of a second wound at the donor site, the three-week delay needed to obtain sufficient amounts of cells, and the absence of a dermal component resulting in low graft take and wound contraction.

Concurrently, allogeneic cell-based engineered skin substitutes have been proposed. Where they offer off-the-shelf temporary wound coverage acting as biologically active dressings releasing growth factors, cytokines and extra cellular matrix components essential for proper wound healing, they are susceptible of immune rejection that is their major weakness Fetal skin, before the third trimester of gestational age, heals rapidly without scar formation conversely to adult skin. Minimal inflammation, specific cytokine and growth factor profiles, and faster and organized deposit and turnover of Extra Cellular Matrix (ECM) components during fetal wound healing have been proposed to explain the absence of scar formation. Because of their low immunogenicity, and their unique regeneration properties, fetal skin cells represent an attractive alternative to the commonly used autologous and allogenic cutaneous grafts.

The investigators developed a new healing dressing constituted by a collagen sponge seeded with a specific ratio of active fetal fibroblasts and keratinocytes producing a variety of wound healing growth factors and cytokines which increase the speed of wound healing, induce an immunotolerant state, with a low inflammatory reaction.

This prospective randomized controlled study aims to compare wound healing of CICAFAST versus conventional treatment (JELONET®) in the treatment of split-thickness skin graft donor site at D8. The patient will be his own control.

ELIGIBILITY:
Inclusion Criteria:

* Female or male aged ≥18 years old
* For potentially childbearing female, only those with effective contraception (contraception pill, implant and intrauterine device) could be included
* Patient who need skin graft ( height equal to or greater than 100cm2 and thickness 1.2mm) after surgery excision
* Patients with social security
* Patients able to understand and follow the trial instructions
* Patients who have signed an informed consent

Exclusion Criteria:

* Patients with an history of cancers except basal and squamous cell, cutaneous carcinoma.
* Patients suffering from uncontrolled metabolic disease (for instance diabete), from a psychiatric disorder not treated, with severe arteritis of lower and/or upper limbs, treated with anticoagulant (unless treatment stops 7 days before the surgery), with severe venous insufficiency, suffering of severe polyneuropathy, with known allergy to antibiotics,
* Patients with an allergic predisposition or known allergy to bovine collagen or silicone
* Patients receiving corticosteroids, immunosuppressive or cytotoxic agents unless treatment stops 4 weeks before the surgery
* Patients contraindicated with local anesthetic used in STSG process of his investigator center
* Patients with systemic infection (all grade defined by CTCAE Common Terminology Criteria for Adverse Event V4.03) at surgery visit will not be included in this trial because of the contraindication of the surgical gesture.
* Patient intolerant to the conventional treatment (JELONET®)
* Patient intolerant to URGO TUL®
* Patient intolerant to TELFA®
* Patient intolerant to the stretchable strip (HYPAFIX® or NYLEX®)
* Pregnant or breast-feeding women
* Patients participating in clinical trial
* Vulnerable people: persons deprived of liberty; under trusteeship or under curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2018-05-16 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
wound healing | Day 8
  The number of complete healing at D8 judged by physician observer. Healing is defined as 80% or more wound closure.

SECONDARY OUTCOMES:
concordance between the healing at D8 (or D11 and D15) judged by physician observer and by another physician using photographs | Day 8 (or D11 and D15 if the healing is not completed)
  The healing at D8 (or D11 or D15 if the healing is not completed) judged by an expert physician on picture. Healing is defined as 80% or more wound closure.
wound healing's rapidity of CICAFAST versus conventional treatment (JELONET®) in the treatment of STSG donor site. | D8 And D11 (if the healing is not completed) and D15 (if the healing is not completed)
  Time to healing (in days) judged by physician observer
tolerance of CICAFAST versus the conventional treatment (JELONET®) | 6 months
  • AE notification: case of infection: patients with grade 1 or 2 infections may be controlled by antibiotherapy. Patients with grade 3 or 4 infection or with biological dressing (CICAFAST) rejection will have CICAFAST dressing removed. However they will stay in the study. Immunological monitoring will be performed to follow a CICAFAST reject of the patient at donor site level.
pain of the wound healing with CICAFAST versus conventional treatment (JELONET®) | Day 8 And D11 (if the healing is not completed) and D15 (if the healing is not completed)
  Number of painful day/wound from the surgery until the complete healing
quality of the wound healing with CICAFAST versus conventional treatment (JELONET®) | 6 months
  Evaluation of the quality of the wound healing by an observer (physician who will not do the patient surgery) at M3 and M6, OSAS (observer scar assessment scale ; 1= normal skin, 10= worst imaginable scar) will be used. By the patient PSAS (patient scar assessment scale ; 1= normal skin, 10= very different) will be used and expertise on picture by 2 external experts (Visual Analogue Scale 10 the worst scar to 1 like normal skin). A second evaluation of complete healing will be performed by two exterior independent experts evaluating the photographs taken until complete healing (Healing is defined as 80% or more wound closure)
quality of the wound healing with CICAFAST versus conventional treatment (JELONET®) for the patient who will have confocal microscopy | 3 months
  Results of scars confocal microscopy at M3

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte Dréno, Pr, Principal Investigator — Nantes University Hospital
Locations (2):
- France (2):
  - Chu de Nantes, Nantes
  - CHU de Nantes, Nantes

REFERENCES:
- [Derived] Poinas A, Perrot P, Lorant J, Nerriere O, Nguyen JM, Saiagh S, Frenard C, Leduc A, Malard O, Espitalier F, Duteille F, Chiffoleau A, Vrignaud F, Khammari A, Dreno B. CICAFAST: comparison of a biological dressing composed of fetal fibroblasts and keratinocytes on a split-thickness skin graft donor site versus a traditional dressing: a randomized controlled trial. Trials. 2019 Oct 28;20(1):612. doi: 10.1186/s13063-019-3718-4. PMID 31661012